CLINICAL TRIAL: NCT07210424
Title: Comparative Study on the Post-operative Pain and Other Outcomes of Mesh Fixation With Prolene vs Vicryl vs Skin Staples in Lichtenstein Inguinal Hernia Repair.
Status: Not yet recruiting | Type: Observational
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 511/RC/KEMU
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Skin Staples: Mesh fixation by skin staples
  Interventions: Procedure: Mesh Fixation
- Sutures: Mesh fixation by sutures (vicryl and prolene)
  Interventions: Procedure: Mesh Fixation

INTERVENTIONS:
Procedure: Mesh Fixation — Mesh fixation during Lichtenstein inguinal hernia repair.

SUMMARY:
We are going to see the outcome measures for patient and compare them across two groups, those who are undergoing mesh fixation for inguinal hernia by sutures, and those who are fixated by skin staples.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing inguinal hernia repair
* 18-65 years
* Both genders

Exclusion Criteria:

* COPD
* Immunocompromised
* Obstructive Uropathy
* Chronic constipation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with inguinal hernia undergoing mesh hernioplasty
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pain | At 3, 7, 14 and 30 post op day
  Pain scores at 3, 7, 14 and 30 days using a Visual Analogue Pain Scale with values ranging between 0 to 10, 0 meaning no pain and 10 being the highest level of pain.

IPD SHARING:
Plan to Share IPD: No